CLINICAL TRIAL: NCT05575687
Title: Brain and Glycemic Responses to Soft Drinks With Different Sweeteners
Brief Title: Brain and Glycemic Responses to Sweet Soft Drinks
Acronym: SWEETBRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Tate & Lyle (Industry)
Responsible Party: Principal Investigator, Paul Smeets, Principal Investigator, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL81742.091.22
Record Dates: First submitted 2022-10-04; First posted 2022-10-12 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Normal Physiological Response to Sweet Drinks
MeSH Terms: interventions — Water; Sucrose; trichlorosucrose; stevioside; psicose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: With the exception of the water treatment, treatment type will be blind for the participants and the researchers. The primary analysis will be performed completely blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Water (Other): Ingestion of 500 ml of mineral water
  Interventions: Other: Water (reference)
- Sucrose (Other): Ingestion of 500 ml of a flavored mineral water sweetened with sucrose
  Interventions: Other: Sucrose
- Sucralose (Other): Ingestion of 500 ml of a flavored mineral water sweetened with sucralose
  Interventions: Other: Sucralose
- Stevia (Other): Ingestion of 500 ml of a flavored mineral water sweetened with stevia extract
  Interventions: Other: Stevia
- Monk fruit (Other): Ingestion of 500 ml of a flavored mineral water sweetened with monk fruit extract
  Interventions: Other: Monk fruit
- Allulose + stevia (Other): Ingestion of 500 ml of a flavored mineral water sweetened with allulose and stevia extract
  Interventions: Other: Allulose + stevia

INTERVENTIONS:
Other: Water (reference) — Ingestion of 500 ml mineral water
  Arms: Water
Other: Sucrose — Ingestion of 500 ml of a flavored mineral water sweetened with sucrose
  Arms: Sucrose
Other: Sucralose — Ingestion of 500 ml of a flavored mineral water sweetened with sucralose
  Arms: Sucralose
Other: Stevia — Ingestion of 500 ml of a flavored mineral water sweetened with stevia extract
  Arms: Stevia
Other: Monk fruit — Ingestion of 500 ml of a flavored mineral water sweetened with monk fruit extract
  Arms: Monk fruit
Other: Allulose + stevia — Ingestion of 500 ml of a flavored mineral water sweetened with allulose and stevia extract
  Arms: Allulose + stevia

SUMMARY:
The goal of this observational study is to determine changes in brain activity and blood sugar in response to the ingestion of flavored waters sweetened with either the nutritive sugar sucrose or different low-caloric sweeteners in healthy normal-weight individuals aged between 18 and 30 years.

The main question it aims to answer is in how far brain and glycemic responses differ between a sugar-sweetened drink and drinks sweetened with different low-caloric sweeteners.

Participants will visit after an overnight fast six times and then have an MRI brain scan before and after consumption of 500 ml of one of the study drinks (beverage sweetened with sucrose or one of four non-caloric sweeteners, or water).

DETAILED DESCRIPTION:
Rationale: The brain is crucial in the regulation of energy intake and maintaining homeostasis which is subserved by an interaction of homeostatic and reward-related brain areas. These brain areas integrate multiple neural and hormonal signals related to energy content such as sweet taste and food reward in the form of ingested energy. Sugar-sweetened soft drinks have been shown to contribute to overconsumption and obesity. Therefore, there is great consumer interest in drinks with low-caloric sweeteners because they do not contribute to energy intake while still providing the hedonic experience of sweet taste. However, different low-caloric sweeteners may have differential effects on the brain because of (subliminal) taste difference and their different metabolic fate. We hypothesize that the brain and glycemic responses to drinks sweetened with sugar and different low-caloric sweeteners will be different. This may have implications for their reward value.

Objective: To determine changes in brain activity in response to the ingestion of flavored waters sweetened with either the nutritive sugar sucrose or different low-caloric sweeteners.

Study design: Randomized crossover design with six treatments. Study population: 30 healthy, non-smoking, normal-weight individuals, aged between 18 and 30 years.

Intervention: Participants will be scanned using MRI before and after consumption of six 500-ml drinks: water; water + sucrose; water + sucralose; water + stevia extract; water + allulose + stevia; water + monk fruit extract. Regional cerebral blood flow (rCBF) and resting state functional MRI (rsfMRI) scans will be made at baseline and at t=5 and t=30 min. Additionally, gastric emptying of the drinks will be examined through gastric MRI at t=15, 25 and 45 min. Blood samples will be collected to measure changes in insulin and glucose levels at baseline and at t=5, 15, 30, 45 and 60 min for all sweet treatments. Participants will rate their appetite and thirst at baseline and at t=15, 25, 30, 45 and 60 min.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years
* BMI between 18.5 and 25 kg/m2
* Apparently healthy (self-reported)
* Right-handed (because brain responses may differ between right- and left handed individuals)
* Sufficient blood hemoglobin (Hb) levels (women > 7,5; men > 8.5 g/dl) and having antecubital veins suitable for blood sampling via a catheter
* Willing to comply with the study procedures
* Willing to be informed about incidental findings of pathology and consenting to informing their general practitioner about this.

Exclusion Criteria:

* Having disturbances of glucose metabolism such as being prediabetic or diabetic
* Use of medication that could influence study results including insulin/metformin/proton pump inhibitors, antacids, anti-depressants
* Allergy or intolerance for any of the study products/compounds (sucrose, sucralose, stevia extract, allulose, monk fruit extract)
* Being a regular smoker (smoking more than one cigarette or e-cigarette with nicotin per day)
* Drinking more than 14 glasses of alcohol a week
* Having genetic, psychiatric or neurological diseases affecting the brain
* Gastric disorders or regular gastric complaints (more than once per week), for example heart burn
* Having renal or hepatic disease
* Using recreational drugs more than once per week (e.g. marihuana, XTC, GHB, laughing gas)
* Having given a blood donation in the past two months
* Being pregnant, lactating or planning on becoming pregnant during the study
* Currently following or having followed calorie-restricted diet in the past two months
* Participating in other research during the study period
* Not having a general practitioner
* Being an employee or student of the Division of Human Nutrition and Health
* Having a contra-indication to MRI scanning

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Local brain perfusion | T=5 and T=30 minutes after the start of consumption
  Change from baseline rCBF in homeostatic and reward-related brain areas in a priori regions of interest (hypothalamus, ventral striatum, dopaminergic midbrain) over time

SECONDARY OUTCOMES:
Seed-based functional connectivity | T=5, T=30 minutes after the start of consumption
  Change from baseline in seed-based functional connectivity of a priori regions of interest (hypothalamus, ventral striatum, dopaminergic midbrain) over time
Blood plasma glucose | T=5, 15, 30, 45 and 60 minutes after the start of consumption
  Change from baseline plasma glucose over time
Blood plasma insulin | T=5, 15, 30, 45 and 60 minutes after the start of consumption
  Change from baseline plasma insulin over time
Gastric content volume | Baseline, T=15, 25 and 45 minutes after the start of consumption
  Change from baseline gastric content volume over time in milliliter as determined from an abdominal MRI scan

OTHER OUTCOMES:
Subjective ratings | T=15, 25, 30, 45 and 60 minutes after the start of consumption
  Verbal subjective ratings of appetite, thirst and wellbeing provided on a scale of 0 - 100 units
Beverage ratings | T=0 minutes (after a few sips)
  Verbal ratings of beverage sweetness and pleasantness on a scale of 0 - 100 units

CONTACTS AND LOCATIONS:
Overall Officials: Paul Smeets, PhD, Principal Investigator — Wageningen University
Locations (1):
- Human Research Unit - Division of Human Nutrition and Health, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: No